CLINICAL TRIAL: NCT02835001
Title: Impact of Reduction Lung Volume Reduction by Coil on Hyperinflation in Severe Emphysema
Brief Title: Hyperinflation Assessment After Treatment by Lung Volume Reduction Coil
Acronym: HEAT-LVRC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change of technique
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/15/7857
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with severe emphysema (Other): Patients with severe emphysema, stable, symptomatic, not controlled despite of international recommendations treatments will have bronchoscopy
  Interventions: Procedure: Bronchoscopy; Device: Lung Volume Reduction Coil (HEAT-LVRC)

INTERVENTIONS:
Procedure: Bronchoscopy — Two sequences of 30 minutes are necessary by patient
Device: Lung Volume Reduction Coil (HEAT-LVRC) — Bronchoscopy with Heat-LVRC

SUMMARY:
Hyperinflation Assessment After Treatment by Lung Volume Reduction Coil (HEAT-LVRC) on Hyperinflation in Severe Emphysema

DETAILED DESCRIPTION:
Two sequences (around 30 minutes) are necessary by patient. Under general anesthesia, two lobs treatment ( 10 Coil by lob) successively introduced by a bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

* Severe emphysema (recent CT-scan (< 6 mois) )
* Age > 35 ans
* Modified Medical Research Council Scale (mMRC) > 2
* Forced expiratory volume in one second (FEV1) post-bronchodilatator < 45%
* Residual volume > 175%
* Total Pulmonary capacity > 100%

Exclusion Criteria:

* Forced expiratory volume in one second (FEV1) variability > 20% after bronchodilatator
* Carbon Monoxide Diffusing Capacity (TLCO) < 20%
* Recurrent respiratory infection Infections with clinics symptoms
* Pulmonary arterial hypertension (PAH) with Pulmonary Arterial Systolic Pressure (PAPS) estimated with echography > 50 mm Hg
* Impossibility to walk more that 140 meter (6 min test)
* Surgery history of volume reduction or pulmonary transplantation
* Broncho-dilatation with clinic symptoms

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Hyperinflation Assessment After Treatment | 3 months
  Assessed by Lung Volume Reduction Coil

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guibert, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Larrey Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No